CLINICAL TRIAL: NCT07346170
Title: A Phase 2 Study of Short Interval Postoperative Stereotactic Body Radiation Therapy (SBRT) After Surgical Intervention for Spine Metastases
Brief Title: Short Interval Postoperative Stereotactic Body Radiation Therapy (SBRT) After Surgical Intervention for Spine Metastases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25721; NCI-2026-00112 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2026-01-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Spine Metastasis; Stereotactic Body Radiation Therapy (SBRT)
MeSH Terms: interventions — Radiosurgery; Magnetic Resonance Spectroscopy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment - Decompression Surgery (Experimental): Participants diagnosed with metastatic spinal cancer who have undergone spinal decompression surgery will receive Stereotactic Body Radiation Therapy (SBRT) after their operation. The radiation dose, ranging from 16 to 40 Gy, will be determined by the radiation oncologist in accordance with expert guidelines. Precise targeting of the treatment area and identification of nearby organs will be achieved using CT and MRI imaging. SBRT will be administered in one to five sessions (1-5 fractions) in either an inpatient setting or a combination of inpatient and outpatient settings. Participants are followed for 1 year after their last treatment. Participants removed from the study for unacceptable treatment or study-related adverse event(s) are followed until resolution or stabilization of all treatment-related adverse events to grade 2 or lower.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Computed Tomography (CT) Simulation; Procedure: Magnetic Resonance Imaging (MRI); Behavioral: Questionnaires
- Treatment - Debulking Surgery (Experimental): Participants diagnosed with metastatic spinal cancer who have undergone spinal debulking surgery will receive SBRT after their operation. The radiation dose, ranging from 16 to 40 Gy, will be determined by the radiation oncologist in accordance with expert guidelines. Precise targeting of the treatment area and identification of nearby organs will be achieved using CT and MRI imaging. SBRT will be administered in one to five sessions (1-5 fractions) in either an inpatient setting or a combination of inpatient and outpatient settings. Participants are followed for 1 year after their last treatment. Participants removed from the study for unacceptable treatment or study-related adverse event(s) are followed until resolution or stabilization of all treatment-related adverse events to grade 2 or lower.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Computed Tomography (CT) Simulation; Procedure: Magnetic Resonance Imaging (MRI); Behavioral: Questionnaires

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Undergo radiation
Procedure: Computed Tomography (CT) Simulation — Undergo imaging
Procedure: Magnetic Resonance Imaging (MRI) — Undergo imaging
Behavioral: Questionnaires — Participant complete health related, quality of life questionnaire (HRQoL)

SUMMARY:
Current guidelines suggest postoperative spine Stereotactic Body Radiation Therapy (SBRT) should be delivered within 2-4 weeks after surgery. This approach is rife with logistical complications that create delays and barriers for patients accessing care. An alternative approach delivers postoperative spine SBRT soon after surgery, starting within a single hospital stay. This study will investigate the effects of short-term postoperative spine SBRT on wound complications in a safety lead-in, then will transition to a phase 2 trial investigating local tumor control.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the local control rate (LC) of treated metastatic sites in patients who undergo surgery for spinal metastasis followed by short interval postoperative spine Stereotactic Body Radiation Therapy (SBRT).

SECONDARY OBJECTIVE:

I. Evaluate the postoperative wound complication rate in participants who undergo surgery for spinal metastasis followed by short-interval postoperative spine SBRT.

II. Determine the radiation toxicity of short-interval postoperative spine SBRT in participants.

III. Determine the progression-free survival (PFS) in participants who undergo surgery for spinal metastasis followed by short-interval postoperative spine SBRT.

IV. Determine the overall survival (OS) in participants who undergo surgery for spinal metastasis followed by short-interval postoperative spine SBRT.

V. Evaluate the quality of life (QoL) of participants who undergo surgery for spinal metastasis followed by short-interval postoperative spine SBRT.

OUTLINE: Participants will received a short interval postoperative SBRT 3-14 days after standard of care surgery for spinal metastases. The SBRT treatment will be delivered up to five sessions in an inpatient or outpatient setting. Participants are follow-up for at month 1, 6, and 12 after SBRT, until removal from study or death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a histologically or cytologically confirmed diagnosis of metastatic malignancy or must have preliminary histology or cytology consistent with a diagnosis of metastatic malignancy.
2. Participants must be considered candidates for postoperative SBRT by the treating radiation oncologist.
3. Participants must have undergone, within the past 13 days, or are planned to undergo minimally invasive or open surgery for the management of a spine metastasis.
4. Disease at any spine level is allowed.
5. Prior therapy

   1. There is no limit on the number of prior spine surgeries or prior courses of radiotherapy directed at the spine if prior therapies occurred at different spinal levels outside the anticipated treatment field.
   2. There is no limit on the number of courses or types of radiotherapy for radiation delivered outside the planned treatment field.
6. Cleared by the primary surgical team for postoperative SBRT, including but not limited to hemodynamic, respiratory, and neurologic stability postoperatively, without immediate postoperative complications noted.
7. Age ≥18 years.
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 70%, see Appendix 1) 1 month prior to presentation for surgery.
9. Estimated survival >3 months or survival considered adequate to undergo spine surgery as assessed by the primary surgical team.
10. Ability to understand and the willingness to sign a written informed consent document.
11. Ability to understand and willingness to comply with treatment schedule, follow-up visits, laboratory testing, and other requirements of the study, including disease assessment by MRI.
12. Individuals with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
13. The effects of radiation on the developing human fetus are generally considered detrimental. Because the radiation therapy used in this trial is known to be teratogenic, individuals of reproductive potential must agree to use adequate contraception (e.g., hormonal or barrier methods, abstinence) for the duration of study participation and for at least 120 days after the last administration of radiation therapy. Should a study participant or their partner become pregnant or suspect pregnancy while participating in this study, they should inform their treating physician immediately.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Prior radiation of any type within the anticipated treatment field (prior radiation outside the anticipated field is acceptable as above).
2. Primary malignancy of the spine (examples: chordoma or sarcoma).
3. Persistent high-grade metastatic spinal cord compression following surgery (Bilsky Grade 3 or higher).
4. Involvement of 3 or more contiguous spinal levels.
5. Involvement of more than 2 non-contiguous spinal levels.
6. American Spinal Injury Association Impairment Scale (ASIA) Grade 3 status.
7. Surgery was a biopsy only.
8. Unable to undergo MRI for any reason.
9. Estimated survival <3 months.
10. Active infection requiring systemic therapy.
11. Active wound complication requiring medical intervention.
12. History of radiation-induced myelopathy from prior spine radiation.
13. History of a collagen vascular disorder (examples: lupus, scleroderma).
14. History of psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. . A woman of childbearing potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Local Control (LC) Rate | 6 months after SBRT
  Local control (LC) is defined as the time from SBRT radiotherapy to metastatic lesions (event) within the SBRT treatment field with stable or decreased size as measured by a board-certified radiologist on follow-up imaging. Participants without any documented events or death will be censored. Estimates and confidence interval will be reported using the Kaplan Meier method.

SECONDARY OUTCOMES:
Median Wound Complication Rate | 1 month after surgery
  Wound complication rate is defined as the rate of participants with wound complications by Centers for Disease Control and Prevention (CDC) criteria. Estimates and the 95% confidence interval will be reported using exact binomial confidence interval (CIs).
Proportion of Participants with Treatment-emergent Adverse Events (TrAE) | 1 month after SBRT
  Proportion of participants with treatment-emergent adverse events as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0) will be reported.
Median Progression-Free Survival (PFS) | Up to 6 months after SBRT
  PFS is defined as the time after enrollment to radiographic progression by RECIST 1.1 criteria on MRI, CT, or Positron Emission Tomography/Computed Tomography (PETCT) at any site of disease, primary or metastatic, or any clinical evidence of progression. Tumor progression is defined as any increase in size within the radiation treatment field (determined by a radiologist), not consistent with or attributable to radiation treatment effect. Hazard ratio and 95% confidence interval will be reported using Kaplan Meier method.
Median Progression-Free Survival (PFS) | Up to 12 months after SBRT
  PFS is defined as the time after enrollment to radiographic progression by RECIST 1.1 criteria on MRI, CT, or PETCT at any site of disease, primary or metastatic, or any clinical evidence of progression. Tumor progression is defined as any increase in size within the radiation treatment field (determined by a radiologist), not consistent with or attributable to radiation treatment effect. Hazard ratio and 95% confidence interval will be reported using Kaplan Meier method.
Median Overall Survival (OS) | Up to 6 months after SBRT
  Overall survival is defined as the time after enrollment to death by any cause. Hazard ratio and 95% confidence interval will be reported using Kaplan Meier method.
Median Overall Survival (OS) | Up to 12 months after SBRT
  Overall survival is defined as the time after enrollment to death by any cause. Hazard ratio and 95% confidence interval will be reported using Kaplan Meier method.
Median Score on the Functional Assessment of Cancer therapy, General- 7 (FACT-G7) at 1 month | 1 month
  The FACT-G7 is a 7-item questionnaire designed to measure general health related quality of life (HRQOL) in cancer patients. Each item response score ranges from 0 (not at all) to 5 (very much). The total score is calculated by taking the sum of the scores x 7 divided by the number of items answered, with a total score range from 0 - 28. The higher the score, the better the HRQOL.
Median score on the FACT-G7 at 6 months | 6 months
  The FACT-G7 is a 7-item questionnaire designed to measure general health related quality of life (HRQOL) in cancer patients. Each item response score ranges from 0 (not at all) to 5 (very much). The total score is calculated by taking the sum of the scores x 7 divided by the number of items answered, with a total score range from 0 - 28. The higher the score, the better the HRQOL.
Median score on the FACT-G7 at 12 months | 12 months
  The FACT-G7 is a 7-item questionnaire designed to measure general health related quality of life (HRQOL) in cancer patients. Each item response score ranges from 0 (not at all) to 5 (very much). The total score is calculated by taking the sum of the scores x 7 divided by the number of items answered, with a total score range from 0 - 28. The higher the score, the better the HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Braunstein, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No